CLINICAL TRIAL: NCT00601926
Title: A Phase II Trial Of Avastin (Bevacizumab) In Patients With Metastatic Papillary Renal Cell Carcinoma
Brief Title: Bevacizumab in Treating Patients With Unresectable or Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor patient accrual. Attempts to open at other sites unsuccessful.
Sponsor: Paul Monk (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Paul Monk, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-06111; NCI-2011-03160 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2008-01-22; First posted 2008-01-28 (Estimated); Results first posted 2015-02-18 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Cancer
Keywords: papillary renal cell carcinoma; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): 15 mg/kg over 90 minutes
  Interventions: Biological: bevacizumab

INTERVENTIONS:
Biological: bevacizumab — 15 mg/kg over 90 minutes every 3 weeks
  Other Names: Avastin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of kidney cancer by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying the side effects and how well bevacizumab works in treating patients with unresectable or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the progression-free survival when bevacizumab is administered to patients with unresectable and/or metastatic papillary renal cell carcinoma.
* To further evaluate the safety of bevacizumab in these patients.

Secondary

* To examine, in a preliminary manner, the response rate to bevacizumab in these patients.
* To collect and store blood and urine samples for future analysis.
* To evaluate overall survival when bevacizumab is administered to these patients.

OUTLINE: Patients receive bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed papillary renal cell carcinoma (RCC)

  * Unresectable and/or metastatic disease
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension and is ≥ 10 mm by spiral CT scan
* No known CNS (central nervous system) disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Life expectancy > 6 months
* ANC (absolute neutrophil count) ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL
* Total bilirubin ≤ 2.0 mg/dL
* AST (aspartate aminotransferase) and ALT (Alanine transaminase) < 3 times normal
* Creatinine clearance > 50 mg/mL
* Calcium < 12 mg/dL (when corrected for level of serum albumin)
* No known HIV infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion criteria:

* Inadequately controlled hypertension (defined as systolic blood pressure [BP] > 150 mm Hg and/or diastolic BP > 100 mm Hg on antihypertensive medications)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association class II-IV congestive heart failure
* Myocardial infarction or unstable angina within the past 6 months
* Stroke or transient ischemic attack within the past 6 months
* Significant vascular disease (e.g., aortic aneurysm or aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Significant traumatic injury within the past 28 days
* Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by either of the following:

  * Urine protein:creatinine (UPC) ratio ≥ 1.0 at screening
  * Urine dipstick for proteinuria ≥ 2+ OR 24-hour urine protein > 1g
* Known hypersensitivity to any component of bevacizumab

PRIOR CONCURRENT THERAPY:

* No prior systemic treatment for metastatic papillary RCC
* At least 4 weeks since prior palliative radiotherapy of painful areas
* More than 28 days since prior major surgical procedure or open biopsy
* No concurrent major surgical procedure
* More than 7 days since prior core biopsy or other minor surgical procedure, excluding placement of a vascular access device
* Concurrent low-dose acetylsalicylic acid (≤ 325 mg/day) allowed in patients at high-risk for arterial thromboembolic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-02; Primary Completion 2011-08 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Monk, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bevacizumab
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) When Bevacizumab is Administered to Patients With Unresectable and/or Metastatic Papillary Renal Cell Carcinoma.
Description: Progression was defined by using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
months | 12 [3 to 25]

2. Primary Outcome: Response Rate to Bevacizumab in This Population.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response, Disappearance of all target lesions; Partial Response, >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease, neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, no occurrence of progression disease for non-target lesions, and no new lesions.
Time Frame: Up to 2 years
Population: Includes patients with Complete response, partial response or stable disease
Measure: Number; unit: patients
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
patients
  Complete Response | 0
  Progressive Disease | 1
  Partial Response | 2
  Stable Disease | 2

3. Secondary Outcome: Safety of Bevacizumab in This Population of Patients
Description: Grade 3 or higher toxicities according to CTCAE version 3.0
Time Frame: Up to 2 years
Measure: Number; unit: toxicities
Arm/Group | Bevacizumab
Number analyzed (Participants) | 5
toxicities | 15

ADVERSE EVENTS:
Time Frame: Adverse events were graded according to NCI CTCAE version 3.0
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=5)
Sudden Death (Cardiac disorders) | 1 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Grade I and Grade III according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Elevated Creatinine (Investigations) | 1 (5) — Grade I and Grade II according to NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Proteinuria (Renal and urinary disorders) | 4 (15) — Grade I, II, III, IV according to NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Hyponatremia (Metabolism and nutrition disorders) | 5 (21) — Grade I and III according to NCI Common Terminology Criteria for Adverse Evens (CTCAE) Version 3.0
Hypertension (Vascular disorders) | 4 (17)
Platelets (Investigations) | 2 (6)
Syncope (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial closed early due to poor patient accrual. Attempts to open this trial at other sites were not successful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes